CLINICAL TRIAL: NCT05369858
Title: A Phase I Mass Balance and Biotransformation Study of [14C]SKLB1028 in Chinese Healthy Male Subjects
Brief Title: A Mass Balance and Biotransformation Study of [14C]SKLB1028 in Chinese Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: CSPC ZhongQi Pharmaceutical Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: HA114-CSP-010
Record Dates: First submitted 2022-05-06; First posted 2022-05-11 (Actual); Last update posted 2022-05-11 (Actual); Status verified 2022-05

CONDITIONS: Healthy Male Subjects
MeSH Terms: interventions — SKLB1028

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- [14C] SKLB1028 (Experimental): Eligible healthy male subjects received a single oral 150 mg (radioactivity of 120µCi) dose of [14C] SKLB1028
  Interventions: Drug: [14C] SKLB1028

INTERVENTIONS:
Drug: [14C] SKLB1028 — A single 150 mg oral dose of [14C] SKLB1028 containing approximately 120 microcurie of [14C] SKLB1028

SUMMARY:
This is a single-centre, open-label, mass balance and biotransformation study in healthy male subjects utilising a single oral dose of [14C] SKLB1028.

ELIGIBILITY:
Inclusion Criteria:

* 1. Chinese male subjects aged 18 to 40 years (inclusive), with normal bowel movements (1~2 times a day).

  2. A minimum body weight of 50 kg and a body mass index ranging from 19 to 26 kg/m^2 (inclusive).

  3. The male subjects with fertility have no child rearing plan or sperm donation plan with their sexual partners during the trial and within one year after taking the drug, and could take reliable contraceptive measures.

  4. Physical examination, vital signs, laboratory (blood routine, blood biochemistry, coagulation function, urine routine, stool routine and occult blood, etc.), 12 lead ECG, chest X-ray and other tests are normal or abnormal without clinical significance.

  5. Fully understand the purpose and requirements of this trial, voluntarily participate in the clinical trial and sign the written informed consent, and can complete the whole trial process according to the test requirements.

Exclusion Criteria:

* 1. Subjects with allergies or allergic diseases, or allergy to test preparations, any of their ingredients and food, or subjects with special dietary requirements, who can not follow the uniform diet.

  2. Inability to swallow oral medications or presence of diseases that affect absorption, distribution, metabolism, or excretion of study medication, as well as the evaluation of drug efficacy and safety, such as hemorrhoids or perianal diseases with regular/ongoing stool blood, habitual constipation or diarrhea, irritable bowel syndrome, inflammatory bowel disease, etc.

  3. History of gastrointestinal ulcer, bleeding, or clinically significant disease, including but not limited to circulatory, endocrine, nervous, digestive, urinary or blood, immune, mental, or metabolic diseases.

  4. Positive hepatitis B surface antigen (HBsAg), hepatitis C virus antibody (HCV Ab), human immunodeficiency virus (HIV) or treponema pallidum antibody results within 1 month prior to dosing.

  5. Use of any drug that inhibits or induces liver drug-metabolizing enzymes (inducers-barbiturates, carbamazepine, phenytoin, rifampicin, dexamethasone, rifabutin, rifapentine, glucocorticoid, omeprazole; inhibitors-SSRI antidepressants, cimetidine, diltiazem, macrolides, verapamil, imidazole antifungals, sedatives and hypnotics, fluoroquinolones, antihistamines, etc.) within 30 days prior to dosing.

  6. Subjects who have used any medication, biological product, Chinese patent medicine, herbal medicine, nutritional supplements or health care products within 14 days prior to the first dose of study medication, or participated in other clinical studies or participated in a clinical study of test preparation within 3 months prior to the first dose of study medication.

  7. Presence of major surgery or incomplete healing of surgical incision, including but not limited to, any surgery with a significant risk of bleeding, prolonged general anesthesia, biopsy or significant traumatic injury within 6 months prior to dosing.

  8. History of needles or blood fainting, or have difficulty in blood collection or cannot tolerate venipuncture for blood collection.

  9. Presence of alcohol abuse or regular use of alcohol within 6 months prior to dosing, i.e. weekly alcohol intake of more than 21 units (One unit is equivalent to 360 mL beer, 45 mL spirits containing 40% alcohol or 150 mL wine) or a positive urine or breath alcohol test at screening.

  10. Smoking more than 10 cigarettes a day. 11. Presence or history of drug abuse or use of soft drugs (e.g. cannabis) within 3 months prior to dosing, or use of hard drugs (such as cocaine, amphetamine, phencyclidine, etc.) within the 3 months prior to dosing, or positive urine test for drugs of abuse at screening.

  12. Habitual consumption of grapefruit juice or excessive drink (>8 cups per day, 1 cup =250 mL) containing caffeine, including coffee, tea.

  13. Workers who need to be exposed to radioactive conditions for a long time; or have radiation exposure (more than 2 chest/abdominal CT, or more than 3 other types of X-ray examinations) within 1 year prior to dosing or participated in clinical studies of radiopharmaceuticals.

  14. Blood loss or donation of one or more units of blood (400 mL) within 3 months prior to the first dose of study medication, or receive blood transfusion within 1 month.

  15. Not suitable for this study as judged by the investigator for any other reason

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2021-08-06 (Actual); Primary Completion 2021-09-04 (Actual); Study Completion 2021-09-11 (Actual)

PRIMARY OUTCOMES:
Cmax | From time zero up to 144 hours post-dose
  Maximum observed plasma concentration
Tmax | From time zero up to 144 hours post-dose
  Time of maximum observed concentration
AUC0-t | From time zero up to 144 hours post-dose
  Area under the plasma concentration time curve from time zero to the last measurable concentration
AUC0-∞ | From time zero up to 144 hours post-dose
  Area under the plasma concentration-time curve from time zero to infinity
Total radioactivity in urine and faces | From time zero up to 240 hours post-dose

SECONDARY OUTCOMES:
Number of subjects with treatment-related adverse events | Up to approximately 14 days after dosing

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Xuhui Central Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No